CLINICAL TRIAL: NCT02336984
Title: A Phase I/II Trial of HER-2/Neu Pulsed DC1 Vaccine Combined With Trastuzumab for Patients With DCIS
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI left Abramson Cancer Center and study never opened at Moffitt Cancer Center.
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 03114
Record Dates: First submitted 2015-01-09; First posted 2015-01-13 (Estimated); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
Keywords: Ductal carcinoma in situ (DCIS)
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Vaccines; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combination Therapy (Experimental): Combination Therapy: HER-2 pulsed DC1 vaccine with trastuzumab and pertuzumab.
  Interventions: Biological: HER-2 pulsed DC1; Drug: trastuzumab; Drug: pertuzumab

INTERVENTIONS:
Biological: HER-2 pulsed DC1 — Vaccine administered weekly, with no more than 4 weeks delay over the course of 6 vaccines.
  Other Names: vaccine
Drug: trastuzumab — The loading dose of Trastuzumab will be 8 mg/kg and the maintenance dose given week 4 will be 6 mg/kg, both standard doses of trastuzumab.
  Other Names: Herceptin
Drug: pertuzumab — Pertuzumab 420 mg IV will be given at the same time as trastuzumab.
  Other Names: Perjeta

SUMMARY:
The purpose of the study is to treat patients with Ductal carcinoma in situ (DCIS) with a combined treatment of DC1 vaccine with Trastuzumab. In this study the investigators will assess the safety and immunogenicity of the combination therapy. The target population is women over 18 years of age and have a diagnosis of DCIS that express HER-2 3 positive. Participants will receive 6 vaccines along with 2 doses of trastuzumab.

This study began at the Abramson Cancer Center of the University of Pennsylvania and will continue at H. Lee Moffitt Cancer Center and Research Institute.

ELIGIBILITY:
Inclusion Criteria:

* Women >= 18 years.
* Ductal carcinoma in situ (DCIS) that express HER-2 3+ on 10% of the DCIS that have not had definitive surgery are diagnosed by core biopsy or NL surgical biopsy with positive margins.
* Patients that are ER+ will take anti-estrogen therapy for treatment of their DCIS during vaccinations.
* Women of childbearing age with a negative pregnancy test documented prior to enrollment.
* Eastern Cooperative Oncology Group (ECOG) Performance Status Score of 0 or 1.
* Women of childbearing potential must agree to use a medically acceptable form of birth control during their participation in the study.
* Have voluntarily signed a written Informed Consent in accordance with institutional policies after its contents have been fully explained to them.

Exclusion Criteria

* Pregnant or lactating.
* Positive for HIV or hepatitis C at baseline by self-report.
* Potential participants with coagulopathies, including thrombocytopenia with platelet count <75,000, INR> 1.5 and partial thromboplastin time > 50 sec
* Major cardiac illness MUGA or ECHO <50% EF.
* Pre-existing medical illnesses or medications which might interfere with the study as determined by Principal Investigator (PI).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-04-04 (Actual); Study Completion 2016-04-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of Related Adverse Events (AEs) | 5 years
  Occurrence of AEs related to study treatment. Adverse Events will be graded according to NCI Common Toxicity Criteria for Adverse Events (CTCAE) V 4.02.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Czerniecki, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania